CLINICAL TRIAL: NCT06876870
Title: MR-Evaluation of Renal Function in Anesthetized Pediatric Patients
Acronym: MERAPED
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MERAPED; 2025-520627-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Renal Blood Flow; Anesthesia; MRI; Renal Oxygenation
Keywords: Renal Blood flow; Anesthesia; Pediatric; MRI
MeSH Terms: interventions — Anesthesia; Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: Patients are randomized to one out of two possible methods of maintenance anesthesia
Who Masked: Outcomes Assessor
Masking Description: The analyzer of the MRI images of renal blood flow, quantifying volumes will be masked from the method of anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): Propofol Maintenance Anesthesia
  Interventions: Drug: Anesthesia Maintenance Agent
- Sevoflurane (Active Comparator): Sevoflurane Maintenance Anesthesia
  Interventions: Drug: Anesthesia Maintenance Agent

INTERVENTIONS:
Drug: Anesthesia Maintenance Agent — Difference in renal blood flow (RBF) between Propofol and Sevoflurane groups. Quantified by specific Multiparametric MRI metrics (e.g., (Renal blood flow by phase contrast imaging) (regional perfusion by Arterial Spin labeling (ASL) and global and regional oxygenation by Blood oxygen dependent signal (BOLD))
  Other Names: Anesthesia; Sevoflurane; Propofol

SUMMARY:
The goal of this study is to investigate the effect of the anesthetic agents sevoflurane or propofol on the blood flow and oxygen delivery to the kidneys.

Pediatric patients who are planned to undergo an MRI scan with generalized anesthesia will be randomized to either IV anesthesia with propofol or inhalation anesthesia with sevoflurane. Both of these anesthetic methods are commonly used for anesthesia on an everyday basis.

In addition to the clinically indicated MRI, Multiparametric MRI will be performed to visualize the effect of the anesthetic agent on renal blood flow, perfusion and oxygenation.

DETAILED DESCRIPTION:
See the study protocol

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients (1 month -14 years of age)
* Indicated for MRI with anesthesia
* ASA (American Society of Anesthesiologists) physical status I-III

Exclusion Criteria:

* Known renal impairment or chronic kidney disease
* Severe cardiac or pulmonary disease
* Allergy to either Propofol or Sevoflurane
* Contraindications to Magnetic Resonance Imaging
* Contraindications to either Propofol or Sevoflurane
* Declined participation or declined consent from patients, parents or guardians
* Ongoing acute kidney injury

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Differences in RBF, as measured by phase contrast imaging with mpMRI, between propofol and sevoflurane anesthesia. | The extra imaging is expected to take 20-30 minutes.
  Multiparametric MRI via phase contrast imaging to quantify renal blood flow, will be standardized to renal area. By quantifying renal blood flow we will be able to evaluate the effects of propofol and sevoflurane on RBF.

SECONDARY OUTCOMES:
Differences in regional renal tissue perfusion, as measured by arterial spin labelling (ASL) with mpMRI, between propofol and sevoflurane anaesthesia | The whole MpMRI will take around 20-30 minutes all together where the primary and secondary outcomes can later be extracted via analysis of the images
  To investigate the effect of Propofol and Sevoflurane on regional tissue perfusion in the renal cortex and medulla.
Differences in regional and global renal oxygenation, as measured by Blood Oxygen Level Dependent (BOLD) signal via mpMRI, between propofol and sevoflurane anaesthesia. | The whole MpMRI will take around 20-30 minutes all together where the primary and secondary outcomes can later be extracted via analysis of the images
  To explore potential differences related to the Sevoflurane or Propofol on regional and global renal oxygenation.
The difference in relation of RBF to systemic non-invasive blood pressure, between propofol and sevoflurane anaesthesia | The entire MpMRI will take around 20-30 minutes all together where the primary and secondary outcomes can later be extracted via analysis of the images
  To investigate how RBF varies in relation to systemic blood pressure in paediatric patients in generalized anaesthesia with propofol or Sevoflurane.
The difference plasma renin concentration, measured by a blood sample, between propofol and sevoflurane anaesthesia | 1 minute
  To explore the effect of Sevoflurane and Propofol on serum Renin concentration as a surrogate marker for Renal sympathetic nerve activation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frithiof, Professor, Study Chair — Istitution of Surgical Sciences, Anesthesiology and Intensive Care

IPD SHARING:
Plan to Share IPD: No
GDPR